CLINICAL TRIAL: NCT06113198
Title: A Phase 4, Single-arm, Open-label, Multi-center Study to Assess the Immune Response and Safety of the Meningococcal Group B Vaccine MenB+OMV NZ When Administered to Healthy Infants From 2 Months of Age in the Republic of Korea
Brief Title: A Study on the Immune Response and Safety of a Vaccine Against N. Meningitidis Serogroup B Infection in Healthy Infants From 2 Months of Age
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 219967
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Meningitis, Meningococcal
Keywords: Neisseria meningitidis; Meningitis; Meningococcal disease; Healthy infants; Safety; Immunogenicity; Republic of Korea
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis; Meningococcal Infections

STUDY DESIGN:
Masking Description: Data will be collected in an open label manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rMenB+OMV NZ Group (Experimental): Participants received rMenB+OMV NZ on Day 1, Day 61, and any day between Day 241- Day 391.
  Interventions: Biological: rMenB+OMV NZ

INTERVENTIONS:
Biological: rMenB+OMV NZ — 3 doses of rMenB+OMV NZ vaccine administered intramuscularly on Day 1, Day 61, and any day between Day 241 - Day 391.

SUMMARY:
The purpose of this study is to assess the safety and immune responses of rMenB+OMV NZ vaccine when administered to healthy infants from 2 months in the Republic of Korea according to a 2-dose primary schedule and 1 booster dose.

DETAILED DESCRIPTION:
As a post-approval commitment to the Ministry of Food and Drug Safety, Bexsero, which is approved in the Republic of Korea for active immunization against MenB, participants will receive a primary series of 2 doses of rMenB+OMV NZ vaccine, with the first dose given at 2 to 5 months of age and the second dose 2 months later. A third dose (booster) will be administered at 12 to 15 months of age. Routine infant vaccines may be administered as per the Korean Routine Immunization Schedule. However, there will be a minimum interval of 14 days before and after the administration of rMenB+OMV NZ vaccine or any other vaccine (21 days for live attenuated vaccines and 7 days for influenza vaccines).

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent(s)/Legally acceptable representative(s) [LAR(s)], who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Healthy participants as established by medical history and clinical examination before entering the study.
* Born full term (i.e., after a gestation period of ≥37 weeks).

Exclusion Criteria:

* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Known exposure from birth to an individual with laboratory confirmed N. meningitidis infection.
* Progressive, unstable or uncontrolled clinical conditions.
* Any contraindications to group B meningococcal vaccine, including but not limited to: history of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Medical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any neuroinflammatory condition (including but not limited to: demyelinating disorders, encephalitis or myelitis of any origin), any congenital neurological condition, encephalopathies, seizures (including all subtypes such as: absence seizures, generalized tonic-clonic seizures, partial complex seizures, partial simple seizures).
* Congenital or peripartum disorders resulting in a chronic illness (including but not limited to: chromosomal abnormalities, cerebral palsy, metabolism or synthesis disorders, cardiac disorders).
* Other serious chronic illness.
* Hypersensitivity to latex.
* Abnormal function of the immune system resulting from clinical conditions, or administration of antineoplastic and immunomodulating agents or radiotherapy for any duration from birth or autoimmune disorders (including, but not limited to: blood, endocrine, hepatic, muscular, nervous system or skin autoimmune disorders) or immunodeficiency syndromes (including, but not limited to: acquired immunodeficiency syndromes and primary immunodeficiency syndromes).
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant Therapy:

* Use of any investigational or non-registered product (drug, vaccine or medical device) since birth, or their planned use during the study period.
* Previous vaccination with any group B meningococcal vaccine at any time prior to informed consent.
* Administration of long acting (defined as administered once per week or less frequently) immunosuppressants, including monoclonal antibodies (e.g., infliximab) since birth and/or planned use at any time during the study period.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) since birth and/or planned use of long-acting immune-modifying treatments at any time during the study period. For corticosteroids, this will mean prednisone equivalent 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products or plasma derivatives since birth and/or planned use at any time during the study period.

Prior/Concurrent Clinical Study Experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other Exclusion Criteria

* Child in care.
* Any immediate dependents, family, or household member of study personnel.

Ages: 2 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-02-23 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with hSBA titers equal to or higher than (≥) Lower Limit of Quantitation (LLOQ) against all MenB indicator strains for the vaccine antigens at Day 91 | At Day 91 (30 days after completion of the primary series)
  The assessed strains are M14459, 96217, NZ98/254 and M13520.
Percentage of participants with hSBA titers equal to or higher than (≥) Lower Limit of Quantitation (LLOQ) against all MenB indicator strains for the vaccine antigens before the third (booster dose) vaccination | At any day between Day 241-391 (before the booster dose)
  The assessed strains are M14459, 96217, NZ98/254 and M13520.
Percentage of participants with hSBA titers equal to or higher than (≥) Lower Limit of Quantitation (LLOQ) against all MenB indicator strains for the vaccine antigens 30 days after the booster dose | At any day between Day 271 - 421 (30 days after the booster dose)
  The assessed strains are M14459, 96217, NZ98/254 and M13520.

SECONDARY OUTCOMES:
Percentage of participants with any unsolicited adverse events (AEs) | Within 30 days after each vaccination and after any vaccination (vaccine administered at Day 1, Day 61, and any day between Day 241 - Day 391)
  An AE is defined as an untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An unsolicited AE (including both serious and nonserious AEs) is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs must have been communicated by participant's parent(s)/Legally acceptable representative(s) who has signed the informed consent.
Percentage of participants with AEs of special interest (AESI), Serious adverse events (SAEs), AEs leading to withdrawal and Medically attended AEs (MAAEs) | From Day 1 to any day between Day 421- Day 571 (throughout the study period)
  AESIs includes seizures: febrile seizure and arthritis. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity. Any AE is defined as untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A MAAE is an AE for which the participant received medical attention including any symptom or illness requiring hospitalization, or an emergency room visit, or visit to/by a healthcare professional.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Junggu
  - GSK Investigational Site, Kyungki-do
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/